CLINICAL TRIAL: NCT05670691
Title: A Prospective, Staged, Exploratory Clinical Study of Combined Multiparametric MRI and PSMA PET/CT for the Evaluation of Patients With High Suspicion of Prostate Cancer for Direct Radical Prostatectomy Without Prostate Biopsy
Brief Title: a Study of Combined mpMRI and PSMA PET/CT for Highly Suspicious Patients Performing Radical Prostatectomy Without Biopsy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ding-Wei Ye, Professor, Fudan University
Other Study IDs: FUSCC RP without biopsy
Record Dates: First submitted 2022-12-18; First posted 2023-01-04 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Prostatic Neoplasms; Prostatectomy; Prostate Biopsy
Keywords: MRI; PSMA PET/CT; prostate biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational, open, single-arm, prospective, staged entry（based on Fleming's Group-Sequential Design） clinical study

The Goal is to evaluate the feasibility and clinical value of direct robot assisted laparoscopic radical prostatectomy without prostate biopsy in patients with high clinical suspicion of prostate cancer based on a prostate MRI PI-RADS score of ≥4 and the PSMA PET/CT positive criteria.

The Primary endpoint is positive pathological diagnosis of prostate cancer after direct radical prostatectomy without prostate biopsy.

The question addressed is whether the feasibility of biopsy-free radical prostatectomy could be scientifically and rationally derived based on Fleming's Group-Sequential design.

DETAILED DESCRIPTION:
Prostate biopsy is currently the key method for diagnosing prostate cancer. However, there are various risks associated with prostate biopsy. First, biopsy complications occur and usually include bleeding, infection, urinary retention, and vasovagal reflexes. Bleeding is one of the most common complications following prostate biopsy, with perineal biopsy hematuria occurring in 39%-44% of cases, rectal bleeding in 17%-27% of cases, and hematospermia in 12%-16% of cases. Infection is one of the more definite complications of prostate biopsy. The incidence is 5-12%. The probability of urinary retention after prostate biopsy is 0.5% to 1.7%. The vasovagal reflex is mainly characterized by a rapid drop in blood pressure, pallor, sweating, nausea, vomiting, chest tightness and, in severe cases, transient coma. The incidence is 0.9% to 16.7%. It is usually necessary to wait 2-4 weeks after biopsy before radical prostate cancer surgery can be performed. Therefore, timely treatment of the patient may be delayed. Second, the pain, anxiety and even fear associated with the biopsy are always with the patient. Third, the issuance of pathology reports generally takes 7-8 days and, if immunohistochemistry is involved, another 2 weeks, a long time with limited management of the full course of the disease, as well as patient attrition.

Multiparametric MRI (mpMRI) has a high tissue resolution and ideal specificity and sensitivity. mpMRI PI-RADS scores of 3, 4 and 5 were associated with a 35%, 60% and 91% diagnosis of prostate cancer, and furthermore, 17%, 34% and 67% diagnosis of CsPCa, respectively.

On the other hand, prostate-specific membrane antigen (PSMA) can specifically anchor prostate cancer cells and has a high sensitivity and specificity for detection.Studies have shown that 68Ga-PSMA PET/CT has a sensitivity of 88%-92% and a specificity of 92%-95% for the diagnosis of prostate cancer. In recent years, PET has also been combined with MRI to obtain many advantages in PET functional imaging as well as MRI imaging discrimination, which is more effective in improving the positive rate of impact diagnosis of prostate cancer.

The combined assessment of multiparametric MRI and PSMA PET/CT has greatly increased the likelihood of prostate cancer in people with multiple abnormalities, and on the other hand, the complications associated with prostate biopsy as well as the delay in surgery and the resulting increased difficulty of surgery. In December 2021, the European Journal of Urology first reported on radical surgery for prostate cancer without biopsy .

The investigators designed this clinical trial based on a combination of multiparametric MRI and PSMA PET/CT to evaluate patients with high suspicion of prostate cancer and make quantitative statistics. mpMRI and PSMA PET/CT were not only among the study parameters, but also could be satisfied with PSMA PET/CT, which was implemented after signing an informed consent after interpretation and performing a direct radical surgery without prostate biopsy.

More importantly, the investigators used Fleming's Group-Sequential Design for the first time, which met the sample size requirements while avoiding the dilemma of having to recruit more patients for the study.

Fleming's Group-Sequential Design

N=71，P0=0.900， P1=0.980 Alpha=0.0230 Power=0.8067

Stage; Sample Size; Cumulative Sample Size; Accept H0 if R ≤ Ag; Reject H0 if R ≥ Rg;

①. 24; 24; 22 27

②. 24; 48; 45 48

③. 23; 71; 68 69

Explanation and description of "Stage Results of Fleming's Group-Sequential Design":

(1) P0=0.900, defined as a pathologically minimum acceptable prostate cancer positivity rate of 90% in the population of patients undergoing biopsy-free radical prostatectomy.

2) P1=0.980, defined as a pathologically desirable prostate cancer positivity rate of 98% in the population of patients undergoing biopsy-free radical prostatectomy.

3) Based on the Fleming group sequential trial design idea, the sample size is calculated using PASS11 software, with 24 cases in the first stage, 24 cases in the second stage, and 23 cases in the third stage, for a total sample size of 71 cases.

5) The protocol is implemented until the completion of the first phase a) If the number of positive cases of pathology after biopsy-free radical prostatectomy is ≤ 22, it indicates the end of this study and concludes that biopsy-free radical prostatectomy is not feasible.

b) If the number of positive cases is 23 or 24, then proceed to the second phase.

6) The protocol is implemented until the completion of the second phase a) If the number of positive cases is ≤45, it indicates the end of this study and concludes that biopsy-free radical prostatectomy is not feasible.

b) If the number of positive cases is 48, it indicates the end of this study and concludes that biopsy-free radical prostatectomy is feasible.

c) If the number of positive cases is 46 or 47, it suggests that the study needs to enter the third phase.

7) Implementation of the protocol to completion of phase III

1. If the number of positive cases is ≤68, this indicates the end of the study and concludes that radical biopsy-free radical prostatectomy is not feasible.
2. If the number of positive cases is ≥69, it indicated the end of the study and concluded that biopsy-free radical prostatectomy is feasible.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years.
2. consent and ability to complete a multiparametric MRI of the prostate.
3. consent and ability to complete PSMA PET/CT.
4. multiparametric MRI of the prostate with a PI-RADS score of 4 or 5 for suspicious lesions.
5. Positive PSMA PET/CT. Its positive is defined as a suspicious lesion score of 2 or 3 (see remarks for specific scoring criteria).
6. good physical condition with an ECOG score of 0 or 1.
7. no history of radiotherapy or other surgery to the pelvis
8. the presence of pelvic lymph node enlargement (>2 cm) or metastasis is allowed; ≤5 bone and lymph node metastases are allowed
9. the patient has good cardiac, pulmonary, hepatic and renal function and is able to tolerate local treatment (surgery or external radiotherapy) of the primary site and metastases, and the treatment will not cause serious complications for the patient.
10. the patient participates voluntarily and has signed an informed consent form
11. the patient is able to receive treatment and subsequent follow-up
12. the expected survival time is greater than 1 year.

Exclusion Criteria:

1. unwillingness or inability to perform multiparametric MRI of the prostate; or PI-RADS score of 0-3
2. request for prostate puncture biopsy.
3. unwillingness or inability to perform PSMA PET/CT; or PSMA PET/CT score of 0 or 1
4. refusing radical prostate cancer surgery, or choosing other primary lesion treatment modalities other than radical prostate cancer surgery
5. poor physical condition that prevents them from tolerating radical prostate cancer surgery
6. More than 5 bone and lymph node metastases, visceral metastases
7. history of combined other malignant tumors (except basal cell carcinoma of the skin or other tumors that have been cured for more than 5 years)
8. other serious medical conditions, such as: unstable heart disease after treatment, myocardial infarction within 6 months prior to treatment, cardiac function class 3-4 (NYHA); uncontrolled hypertension (>150/90 mmHg, severe neurological or psychological disorders including dementia or epilepsy) with medical treatment; uncontrolled active infection; acute gastric ulcer; hypercalcemia; chronic obstructive lung disease.
9. have participated in other clinical studies prior to enrollment.

Note: Positive PSMA PET/CT, defined as based on the miPSMA score scale suggested by the PROMISE Institute (score 0 - below the depth of blood contrast; score 1 - equal to or above the blood contrast and below the liver contrast; score 2 - equal to or above the liver contrast and below the parotid contrast; score 3 - equal to or above the liver parotid contrast.)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Robotic-assisted laparoscopic radical prostate cancer surgery is recommended for this group of patients. Ultimately, the presence or absence of evidence of malignant prostate cancer on the pathology report after radical prostatectomy is used as an observational endpoint in this study. Relevant perioperative clinicopathological data are also collected according to the study objectives.
Sampling Method: Probability Sample
Enrollment: 71 (Estimated)
Dates: Start 2023-01-10 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
The positive rate of pathological diagnosis of prostate cancer | two years
  The positive rate of pathological diagnosis of prostate cancer from tissue of prostatectomy for the all the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, Doctor, Study Director — Fudan University

IPD SHARING:
Plan to Share IPD: No
The investigators do not provide IPD sharing to other researchers, but do further analysis in this center.

REFERENCES:
- [Result] Meissner VH, Rauscher I, Schwamborn K, Neumann J, Miller G, Weber W, Gschwend JE, Eiber M, Heck MM. Radical Prostatectomy Without Prior Biopsy Following Multiparametric Magnetic Resonance Imaging and Prostate-specific Membrane Antigen Positron Emission Tomography. Eur Urol. 2022 Aug;82(2):156-160. doi: 10.1016/j.eururo.2021.11.019. Epub 2021 Dec 6. PMID 34887117
- [Result] Emmett L, Buteau J, Papa N, Moon D, Thompson J, Roberts MJ, Rasiah K, Pattison DA, Yaxley J, Thomas P, Hutton AC, Agrawal S, Amin A, Blazevski A, Chalasani V, Ho B, Nguyen A, Liu V, Lee J, Sheehan-Dare G, Kooner R, Coughlin G, Chan L, Cusick T, Namdarian B, Kapoor J, Alghazo O, Woo HH, Lawrentschuk N, Murphy D, Hofman MS, Stricker P. The Additive Diagnostic Value of Prostate-specific Membrane Antigen Positron Emission Tomography Computed Tomography to Multiparametric Magnetic Resonance Imaging Triage in the Diagnosis of Prostate Cancer (PRIMARY): A Prospective Multicentre Study. Eur Urol. 2021 Dec;80(6):682-689. doi: 10.1016/j.eururo.2021.08.002. Epub 2021 Aug 28. PMID 34465492
- [Result] Chen M, Zhang Q, Zhang C, Zhou YH, Zhao X, Fu Y, Gao J, Zhang B, Wang F, Qiu X, Guo H. Comparison of 68Ga-prostate-specific membrane antigen (PSMA) positron emission tomography/computed tomography (PET/CT) and multi-parametric magnetic resonance imaging (MRI) in the evaluation of tumor extension of primary prostate cancer. Transl Androl Urol. 2020 Apr;9(2):382-390. doi: 10.21037/tau.2020.03.06. PMID 32420143
- [Result] Yang FY, Li YJ, Han SJ, Chen D, Wu LY, Xiao ZJ, Li CL, Xing NZ. [The preliminary clinical study on radical prostatectomy without preoperative prostate biopsy]. Zhonghua Yi Xue Za Zhi. 2020 Sep 15;100(34):2658-2662. doi: 10.3760/cma.j.cn112137-20200104-00021. Chinese. PMID 32921013
- [Result] Moldovan PC, Van den Broeck T, Sylvester R, Marconi L, Bellmunt J, van den Bergh RCN, Bolla M, Briers E, Cumberbatch MG, Fossati N, Gross T, Henry AM, Joniau S, van der Kwast TH, Matveev VB, van der Poel HG, De Santis M, Schoots IG, Wiegel T, Yuan CY, Cornford P, Mottet N, Lam TB, Rouviere O. What Is the Negative Predictive Value of Multiparametric Magnetic Resonance Imaging in Excluding Prostate Cancer at Biopsy? A Systematic Review and Meta-analysis from the European Association of Urology Prostate Cancer Guidelines Panel. Eur Urol. 2017 Aug;72(2):250-266. doi: 10.1016/j.eururo.2017.02.026. Epub 2017 Mar 21. PMID 28336078
- [Result] Eiber M, Weirich G, Holzapfel K, Souvatzoglou M, Haller B, Rauscher I, Beer AJ, Wester HJ, Gschwend J, Schwaiger M, Maurer T. Simultaneous 68Ga-PSMA HBED-CC PET/MRI Improves the Localization of Primary Prostate Cancer. Eur Urol. 2016 Nov;70(5):829-836. doi: 10.1016/j.eururo.2015.12.053. Epub 2016 Jan 18. PMID 26795686